CLINICAL TRIAL: NCT05491785
Title: Randomized, Double-blind, Four Period, Six-treatment, Double-dummy, Placebo Controlled, Partial-crossover Study to Explore and Compare the Ventilatory Response to Hypercapnia (VRH) of Cebranopadol, Oxycodone, and Placebo in Healthy Subjects
Brief Title: Cebranopadol Effects on Ventilatory Drive, Central Nervous System (CNS) and Pain.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PARK-104-VRH
Record Dates: First submitted 2022-07-27; First posted 2022-08-08 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Pain
Keywords: cebranopadol; pain; respiratory; hypercapnia
MeSH Terms: conditions — Pain; Hypercapnia | interventions — 6'-fluoro-4',9'-dihydro-N,N-dimethyl-4-phenylspiro(cyclohexane-1,1'(3'H)-pyrano(3,4-b)indol)-4-amine; Oxycodone

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, four- period, six-treatment, double-dummy, placebo controlled, partial-crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-dummy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cebranopadol 600 µg (Experimental): 3 x 200 µg cebranopadol tablets
  Interventions: Drug: Cebranopadol 600 µg
- Cebranopadol 800 µg (Experimental): 4 x 200 µg cebranopadol tablets
  Interventions: Drug: Cebranopadol 800 µg
- Cebranopadol 1000 µg (Experimental): 5 x 200 µg cebranopadol tablets
  Interventions: Drug: Cebranopadol 1000 µg
- Oxycodone 30 mg (Active Comparator): 3 x 10 mg Oxycodone tablets
  Interventions: Drug: Oxycodone 30 mg
- Oxycodone 60 mg (Active Comparator): 3 x 20 mg Oxycodone tablets
  Interventions: Drug: Oxycodone 60 mg
- Cebranopadol placebo tablets/ Oxycodone placebo capsules (Placebo Comparator): Cebranopadol placebo tablets/ Oxycodone placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cebranopadol 600 µg — Participants will be administered a single dose of 8 identically appearing capsules containing: 3 oxycodone placebo capsules, 3 cebranopadol 200 µg tablets and 2 cebranopadol placebo tablets
  Other Names: Experimental
  Arms: Cebranopadol 600 µg
Drug: Cebranopadol 800 µg — Participants will be administered a single dose of 8 identically appearing capsules containing: 3 oxycodone placebo capsules, 4 cebranopadol 200 µg tablets and 1 cebranopadol placebo tablet
  Other Names: Experimental
  Arms: Cebranopadol 800 µg
Drug: Cebranopadol 1000 µg — Participants will be administered a single dose of 8 identically appearing capsules containing: 3 oxycodone placebo capsules, and 5 cebranopadol 200 µg tablets
  Other Names: Experimental
  Arms: Cebranopadol 1000 µg
Drug: Oxycodone 30 mg — Participants will be administered a single dose of 8 identically appearing capsules containing: 3 oxycodone 10 mg capsules, and 5 cebranopadol placebo tablets
  Other Names: Active Comparator
  Arms: Oxycodone 30 mg
Drug: Oxycodone 60 mg — Participants will be administered a single dose of 8 identically appearing capsules containing: 3 oxycodone 20 mg capsules, and 5 cebranopadol placebo tablets
  Other Names: Active Comparator
  Arms: Oxycodone 60 mg
Drug: Placebo — Participants will be administered a single dose of 8 identically appearing capsules containing: 3 oxycodone placebo capsules, and 5 cebranopadol placebo tablets
  Other Names: Placebo comparator
  Arms: Cebranopadol placebo tablets/ Oxycodone placebo capsules

SUMMARY:
Opioids are potent painkillers but come with serious adverse effects ranging from addiction to potentially lethal respiratory depression via activation of μ-opioid receptors (MOP) at specific sites in the central nervous system. Cebranopadol is a first-in-class investigational drug to treat patients with acute and chronic pain. The molecule dually activates the Nociceptin/Orphanin FQ peptide (NOP) receptor and the classical MOP receptor. This is a unique mechanism of action and has demonstrated efficacy in multiple Phase 2 and Phase 3 clinical studies across several nociceptive and neuropathic indications as well as a superior safety profile, low potential for abuse and minimal risk of physical dependence. In animal studies, cebranopadol produced considerably less respiratory depression at comparably analgesic doses of oxycodone and fentanyl and appeared to have a ceiling to its respiratory effects. Preliminary clinical trials have suggested that these results will be similar in humans.

The present study is designed to investigate if: 1) cebranopadol produces less respiratory depression than oxycodone 2) cebranopadol respiratory effects have a ceiling at very high doses and 3) cebranopadol does not produce significant respiratory depression, as measured in this study design with 30 subjects, at any dose in the VRH model.

DETAILED DESCRIPTION:
This is a randomized, double blind, four period, six-treatment, double-dummy, placebo controlled, partial-crossover study will investigate the effects of cebranopadol on the ventilatory response to hypercapnia (VRH), nociceptive thresholds and safety.

VRH testing is non-invasive and is an established technique to evaluate respiratory depression following the administration of opioids.

The test will be performed using a rebreathing setup with the subjects comfortably seated or semi-supine in a hospital bed and breathing through a facemask. VRH will be performed at several timepoints post-administration of cebranopadol, oxycodone or placebo in a randomized fashion. At each time point, subjects will be allowed an acclimation period of ambient air to establish regular breathing pattern; immediately followed by rebreathing a hypercapnic gas mixture (7%CO2, in oxygen (50%)), for at least 3 min. Between timepoints, subjects will remove their face masks and breathe ambient air.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-mandated procedure.
2. Subject is able to speak, read, and understand Dutch and voluntarily provide written informed consent to participate in the study.
3. Adult men or women aged 18 to 45 years, inclusive.
4. Subjects are in good health as indicated by medical history, physical examination, vital signs, oxygen saturation, clinical laboratory tests, and 12-lead ECG.
5. Body mass index between 18.0 kg/m2 and 32.0 kg/m2 and body weight greater than 50 kg, inclusive.
6. Adequate contraception is being used or women of nonchildbearing potential may be enrolled if surgically sterile (i.e., after hysterectomy) or postmenopausal for at least 2 years (based on subject's report).

Exclusion Criteria:

1. History or presence of clinically significant cardiovascular (incl. a history of risk factors for torsade de pointes e.g., heart failure, hypokalaemia, family history of long QT syndrome, history of myocardial infarction, ischaemic heart disease, clinically significant arrhythmia or uncontrolled arrhythmia or cardiac failure), pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease (e.g., anxiety); or any other condition (e.g., hyperventilation disorder), which, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
2. History of known difficult airway access or uncontrolled gastroesophageal reflux disease (GERD), gastric motility disorders, or delayed gastric emptying
3. Has clinically significant abnormalities on ECG at screening or Day -1, as defined by the following:

   1. prolonged corrected QT interval (Fridericia-corrected QT interval [QTcF] >450 ms in males and >470 ms in females) demonstrated on ECG;
   2. Left bundle branch block at Screening or Baseline
4. Systolic blood pressure (BP) >150 or <90 mmHg or diastolic BP >90 or <50 mmHg at Screening or Baseline, or history of clinically significant orthostatic hypotension.
5. Heart rate (HR) <40 beats per minute (bpm) or >100 bpm at Screening.
6. Is currently enrolled in another clinical study or used any investigational drug or device within 3 months prior to dosing or has participated in more than 4 investigational drug studies within 1 year prior to Screening.
7. Has any condition in which an opioid is contraindicated (e.g., significant respiratory depression, acute or severe bronchial asthma or hypercarbia, or has or is suspected of having paralytic ileus).
8. Have a history of chronic obstructive pulmonary disease or any other lung disease (e.g., asthma, bronchitis, obstructive sleep apnoea, exercise-induced asthma) that would cause CO2 retention.
9. History of opioid use disorder per Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) classification, or other drug/substance or alcohol dependency or abuse (excluding nicotine and caffeine) within the last 5 years before Screening.
10. Has a positive alcohol test or urine drug screen for drugs of abuse (amphetamines, methamphetamines, barbiturates, benzodiazepines, cocaine, and opioids) at Screening or Day -1.
11. Use of nicotine-containing products within 4 weeks before the Screening visit and not able to withhold from smoking during the study.
12. Pregnant or breastfeeding.
13. Subjects indicating pain test intolerability at Screening or achieving pain tolerance at >80% of maximum input intensity for the pain tests.
14. Demonstrated allergic reactions (e.g., food, drug, atopic reactions, or asthmatic episodes) which, in the opinion of the Investigator, interfere with the subject's ability to participate in the trial.
15. Positive hepatitis B surface antigen (HBsAg), hepatitis B core antibodies (Anti-HBc), hepatitis C antibodies (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at Screening.
16. Use of prescription, non-prescription medications or herbal preparations containing St. John's Wort, within 14 days or 5 half-lives prior to dosing, whichever is longer. An exception is made for contraceptives and incidental use of paracetamol or ibuprofen, which is allowed up to 48 hours before start of each visit. Other exceptions are allowed only when clearly documented by the investigator.
17. No vitamin, mineral, herbal, and dietary supplements will be permitted within 7 days prior to study drug administrations, or less than 5 half-lives (whichever is longer, and during the course of the study.
18. Any clinically significant lifetime history of suicidal behaviour or ideation and/or poses a current (within the past 12 months) suicide risk, as assessed by scores on the Columbia Suicide Severity Rating Scale (C-SSRS) at Screening per Investigator judgment
19. Receipt of blood products within 4 weeks, blood donation or blood loss >250 mL within 8 weeks, or donation of plasma within 1 week of any Study Drug dose administration.
20. Is employed by Tris, Park, the Centre for Human Drug Research (CHDR), or the Investigator or study site (permanent, temporary contract worker, or designee responsible for the conduct of the study), or is immediate family* of a Tris, Park, CHDR, Investigator, or study site employee.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Ventilatory response to hypercapnia (VRH) by maximum decrease in minute ventilation (L) | 24 hours
  Pre-dose to 24 h postdose

SECONDARY OUTCOMES:
Pupil constriction compared to baseline (mm) | 24 hours
  Pre-dose to 24 h postdose
Electrical and pressure pain tests | 24 hours
  Pre-dose to 24 h postdose
Adverse event reporting | 24 hours
  Pre-dose to 24 h postdose

CONTACTS AND LOCATIONS:
Overall Officials: Albert Dahan, MD, PhD, Principal Investigator — LUMC; Geert Jan Groeneveld, MD, PhD, Principal Investigator — CHDR
Locations (2):
- Netherlands (2):
  - Centre for Human Drug Research (CHDR), Leiden
  - Leiden University Medical Centre (LUMC), Leiden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dahan A, Boom M, Sarton E, Hay J, Groeneveld GJ, Neukirchen M, Bothmer J, Aarts L, Olofsen E. Respiratory Effects of the Nociceptin/Orphanin FQ Peptide and Opioid Receptor Agonist, Cebranopadol, in Healthy Human Volunteers. Anesthesiology. 2017 Apr;126(4):697-707. doi: 10.1097/ALN.0000000000001529. PMID 28291085